CLINICAL TRIAL: NCT06212791
Title: EXCLAMATORY: EXercise Cardiac Magnetic Resonance Assessment of Left Atrial Mechanics Following Ablation TO Reduce Atrial Fibrillation Burden and Correlation With Exercise CapacitY Longitudinal Study
Brief Title: EXercise Cardiac Magnetic Resonance Assessment of Left Atrial Mechanics Following Ablation
Acronym: EXCLAMATORY
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HM20027087; K23HL166956 (NIH)
Record Dates: First submitted 2023-12-19; First posted 2024-01-19 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Catheter ablation; Exercise capacity
MeSH Terms: conditions — Atrial Fibrillation | interventions — Exercise Test; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients under going catheter ablation: Patients undergoing catheter ablation for paroxysmal AF, reduction or elimination of arrhythmia burden
  Interventions: Behavioral: Self- Report Evaluation-Duke Activity Status Index; Behavioral: Self- Report Evaluation Atrial Fibrillation Effect on Quality of Life Questionnaire; Diagnostic Test: Cardiopulmonary exercise test (CPET); Diagnostic Test: Transthoracic echocardiogram; Diagnostic Test: Ambulatory cardiac rhythm assessment; Diagnostic Test: Cardiovascular magnetic resonance (CMR)

INTERVENTIONS:
Behavioral: Self- Report Evaluation-Duke Activity Status Index — Complete the Self- Report Evaluation-Duke Activity Status Index
Behavioral: Self- Report Evaluation Atrial Fibrillation Effect on Quality of Life Questionnaire — Complete the Self- Report Evaluation, Atrial Fibrillation Effect on Quality of Life Questionnaire
Diagnostic Test: Cardiopulmonary exercise test (CPET) — Cardiopulmonary exercise test (CPET)
Diagnostic Test: Transthoracic echocardiogram — Transthoracic echocardiogram at rest and immediately following peak exercise during CPET
Diagnostic Test: Ambulatory cardiac rhythm assessment — Ambulatory cardiac rhythm assessment
Diagnostic Test: Cardiovascular magnetic resonance (CMR) — Cardiovascular magnetic resonance (CMR) study at rest and during two stages of submaximal exercise (ExeCMR)

SUMMARY:
Longitudinal, observational cohort study to evaluate changes in left atrial (LA) reservoir function during exercise and overall exertional capacity in patients following catheter ablation for paroxysmal atrial fibrillation (AF).

DETAILED DESCRIPTION:
EXCLAMATORY is a longitudinal observational cohort clinical research study to evaluate the effects of catheter ablation for paroxysmal atrial fibrillation on left atrial and left ventricular performance during exercise, as well as effects on overall exercise capacity

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of paroxysmal AF
* Left ventricular ejection fraction ≥50%
* Scheduled for catheter ablation
* Able to speak, hear, and read English
* Willing and able to provide informed consent

Exclusion Criteria:

* Persistent or permanent AF
* Prior ablation (catheter based or surgical) for AF
* Significant sinus node dysfunction
* Implanted pacemaker or defibrillator
* Contraindication to or inability to complete cardiovascular magnetic resonance study
* Contraindication to or inability to complete exercise testing
* Chronic kidney disease with estimated glomerular filtration rate <30 mL/min/1.73m2
* Severe left ventricular hypertrophy
* Unrelated cardiomyopathy that is expected to limit exercise capacity, including but not limited to:

  * Hypertrophic cardiomyopathy
  * Cardiac amyloidosis
  * Constrictive pericarditis
* Pulmonary arterial hypertension
* Prior cardiac surgery
* Active pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In patients undergoing catheter ablation for paroxysmal AF, reduction or elimination of arrhythmia burden will result in favorable LA reverse remodeling - which will result in improved LA reservoir function reserve during exercise, thereby augmenting LV stroke volume reserve during exercise.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in LA reservoir function reserve at submaximal exercise after catheter ablation in patients with paroxysmal AF. | Baseline and the follow up testing will be performed 5-6 months (to be more specific: 150-180 days) after catheter ablation.
  Change in LA reservoir volume reserve from baseline to follow up, change in left ventricular (LV) stroke volume reserve from baseline to follow up, correlation between changes in LA reservoir volume reserve and changes in LV stroke volume reserve. Therefore the follow up testing will be performed 5-6 months (to be more specific: 150-180 days) after catheter ablation.

SECONDARY OUTCOMES:
Change in LV stroke volume reserve at submaximal exercise after catheter ablation in patients with paroxysmal AF. | Baseline and the follow up testing will be performed 5-6 months (to be more specific: 150-180 days) after catheter ablation.
  Change in LA reservoir volume reserve from baseline to follow up, change in LV stroke volume reserve from baseline to follow up, correlation between changes in LA reservoir volume reserve and changes in LV stroke volume reserve.
Correlation between changes in LA reservoir volume reserve and changes in LV stroke vol reserve after catheter ablation in patients with paroxysmal AF | Baseline and the follow up testing will be performed 5-6 months (to be more specific: 150-180 days) after catheter ablation.
  Correlation between changes in LA reservoir volume reserve and changes in LV stroke volume reserve after catheter ablation in patients with paroxysmal AF
Correlation between changes in LA reservoir function reserve at submaximal exercise and changes in mixed venous oxygen tension (pVO2) . | Baseline and the follow up testing will be performed 5-6 months (to be more specific: 150-180 days) after catheter ablation.
  Correlation between changes in LA reservoir function reserve at submaximal exercise and changes in pVO2 after catheter ablation
Correlation between changes in LV stroke volume reserve at submaximal exercise and changes in pVO2 | Baseline and the follow up testing will be performed 5-6 months (to be more specific: 150-180 days) after catheter ablation.
  Correlation between changes in LV stroke volume reserve at submaximal exercise and changes in pVO2 after catheter ablation.
Correlation between baseline AF burden and LA function, LV Function and pVO2 | Baseline and the follow up testing will be performed 5-6 months (to be more specific: 150-180 days) after catheter ablation.
  Correlation between baseline AF burden and LA function (rest and exercise), LV function (rest and exercise), and pVO2
Correlation between the amount of AF burden reduction and the changes in LA function, LV function (rest and exercise), and pVO2. | Baseline and the follow up testing will be performed 5-6 months (to be more specific: 150-180 days) after catheter ablation.
  Correlation between the amount of AF burden reduction and the changes in LA function (rest and exercise), LV function (rest and exercise), and pVO2.

CONTACTS AND LOCATIONS:
Overall Officials: Cory Trankle, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States